CLINICAL TRIAL: NCT05525975
Title: The Impact of Pre-operative Opioid Education and Opioid Disposal Following Shoulder Arthroplasty
Brief Title: Opioid Consumption and Disposal After Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brendan M. Patterson (Other)
Responsible Party: Sponsor-Investigator, Brendan M. Patterson, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202202119
Record Dates: First submitted 2022-08-15; First posted 2022-09-02 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use
Keywords: opioid; Shoulder Arthroplasty; Shoulder Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control/Standard of Care (No Intervention): This arm will follow the standard of care practices of the Shoulder Surgery Department at UIHC, and will work as a control group.
- Education Arm (Experimental): Participants in this arm will receive at their preoperative work-up visit a brochure and will watch an educational video. Both educational materials (brochure and video) will address information about opioid medications, pain management techniques and properly disposal of any excess opioid medication. In addition, participants receive an envelope in which they will be able to dispose their unused opioid pills. These envelopes will be the same ones used in our pilot study (IRB# 202012142). The disposal method consists of secured, labeled envelopes to dispose of the excess of Opioid medication. These envelopes will be provided by "Sharps Compliance, Inc.", a company that manages pharmaceutical waste disposal programs for healthcare facilities. Through their "TakeAway Medication Recovery System Envelope (USPS)" they allow the collection and disposal of controlled substances (Schedules II-IV) and non-controlled medications.
  Interventions: Other: Educational materials

INTERVENTIONS:
Other: Educational materials — Educational materials will be developed by our interdisciplinary research team. Will consist of a brochure and a video. Both materials highlight important information about opioid medications, explain proper disposal of excess of opioid medications and provide drug-free pain management tools for postoperative pain.
  Arms: Education Arm

SUMMARY:
Opioid medications are widely used after many orthopedic procedures and are routinely prescribed after shoulder replacement surgery. Despite the high prevalence of opioid abuse and misuse, there is no standardized mechanism for patients to dispose of unused opioid medications safely and securely and the average number of opioid pills required after shoulder replacement surgery is still unknown. In a prior pilot study conducted by our group (IRB# 202012142), opioid consumption patterns of patients undergoing shoulder arthroplasty were analyzed, as well as their adherence to a safe and secure disposal mechanism for excess opioid pills. A 94% retention rate was achieved and preliminary results showed that most of the subjects were 60 years of age and older.

The objective of the current proposal is to: (1) develop pre-operative education materials related to post-operative opioid use following shoulder arthroplasty; (2) pilot the impact of this educational intervention; (3) examine the effect of providing disposal mechanisms for unused opioid pain medications following shoulder arthroplasty. The proposal is to conduct a single blinded randomized controlled trial of patients undergoing total shoulder replacement, both anatomic total shoulder arthroplasty (TSA) and reverse shoulder arthroplasty (RSA), and Hemiarthroplasty at UIHC. This randomized controlled trial will compare: (1) education plus opioid disposal to the standard of care (SC). The investigators hypothesize that pre-operative opioid education modules combined with a structured opioid disposal program will decrease opioid consumption following shoulder arthroplasty.

DETAILED DESCRIPTION:
Patients will be identified as potential research subjects by one of the the two Shoulder Surgeons (BMP, JVN) during their visit to the Shoulder Surgery Clinic at University of Iowa Hospitals and Clinics, according to the indication of a shoulder arthroplasty.

During their preoperative work-up visit, patients will be invited to participate in the research study. The research coordinator will discuss the study with potential subjects in a private office or exam room. If the patient shows interest in participating, the research coordinator and the patient will go through the process of consent of participants.

After agreeing to participate and signing informed consent, participants will be randomized into one of the 2 study arms at their preoperative work-up visit.

Participants in Arm 1 (control group) will go through all procedures before and after their surgery as they usually do in standard of care practice, and all procedures will continue as scheduled. The standard of care practice of the Shoulder Surgery department at UIHC is that for patients that will undergo a surgical procedure NOT to receive any type of education on Opioid consumption, disposal or risks prior to the surgery.

Participants in Arm 2 (education + disposal), at their work-up visit, will receive a brochure, will watch an educational video, and will also receive an envelope in which they will be able to dispose their unused opioid pills. These envelopes will be the same ones used in the team's previous pilot study (IRB# 202012142). The disposal method consists of secured, labeled envelopes to dispose of the excess of Opioid medication. These envelopes will be provided by "Sharps Compliance, Inc.", a company that manages pharmaceutical waste disposal programs for healthcare facilities. Through their "TakeAway Medication Recovery System Envelope (USPS)" they allow the collection and disposal of controlled substances (Schedules II-IV) and non-controlled medications. Subjects will be explained how to use the envelope and that since it is labeled they will not have to pay for anything when using it. The brochure will address opioid risks, side effects, disposal and explain non-opioid pain management strategies. The educational video will consist of a short video to educate patients on the current opioid crisis, explain how to safely dispose of excess opioids and will teach them about drug-free pain management techniques.

All participants (Arm 1 and Arm2), after their surgery and after being discharged from the hospital, will receive daily text messages with a link to a REDCap survey. This texts will be delivered during the first 2 weeks following surgery. The survey will assess postoperative pain in the last 24 hours through Pain VAS, number of pills taken during the last 24 hours, number of pills disposed, method for disposal.

For participants who did not answer the daily survey and for the ones who are still taking opioids after 2 weeks following surgery, will be able to answer the survey at their postoperative appointment at Shoulder Surgery clinic (2-weeks postop or 6-weeks postop).

Patients in the education group will be emailed after their 6 week post-op visit to inquire as to their overall satisfaction with the education module and post-op buddy app/text program.

Disposal envelops will be tracked via tracking number just to confirm they were received by the disposal center (Sharps Compliance Inc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at UIHC Shoulder Surgery Clinic that are indicated for primary total shoulder arthroplasty procedures.

Exclusion Criteria:

* revision shoulder arthroplasty
* arthroplasty for proximal humerus fractures
* patients with a history of chronic opioid consumption
* patients with contraindications for opioid consumption.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan M Patterson, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Bettlach CLR, Hasak JM, Santosa KB, Larson EL, Tung TH, Fox IK, Moore AM, Mackinnon SE. A Simple Brochure Improves Disposal of Unused Opioids: An Observational Cross-Sectional Study. Hand (N Y). 2022 Jan;17(1):170-176. doi: 10.1177/1558944720959898. Epub 2020 Oct 7. PMID 33025827
- [Background] Lewis ET, Cucciare MA, Trafton JA. What do patients do with unused opioid medications? Clin J Pain. 2014 Aug;30(8):654-62. doi: 10.1097/01.ajp.0000435447.96642.f4. PMID 24281287
- [Background] Kumar K, Gulotta LV, Dines JS, Allen AA, Cheng J, Fields KG, YaDeau JT, Wu CL. Unused Opioid Pills After Outpatient Shoulder Surgeries Given Current Perioperative Prescribing Habits. Am J Sports Med. 2017 Mar;45(3):636-641. doi: 10.1177/0363546517693665. Epub 2017 Feb 9. PMID 28182507
- [Background] Saunders KW, Dunn KM, Merrill JO, Sullivan M, Weisner C, Braden JB, Psaty BM, Von Korff M. Relationship of opioid use and dosage levels to fractures in older chronic pain patients. J Gen Intern Med. 2010 Apr;25(4):310-5. doi: 10.1007/s11606-009-1218-z. Epub 2010 Jan 5. PMID 20049546
- [Background] Sabesan VJ, Stankard M, Grauer J, Echeverry N, Chatha K. Predictors and prescribing patterns of opioid medications surrounding reverse shoulder arthroplasty. JSES Int. 2020 Oct 9;4(4):969-974. doi: 10.1016/j.jseint.2020.08.014. eCollection 2020 Dec. PMID 33345242
- [Background] Martusiewicz A, Khan AZ, Chamberlain AM, Keener JD, Aleem AW. Outpatient narcotic consumption following total shoulder arthroplasty. JSES Int. 2020 Jan 16;4(1):100-104. doi: 10.1016/j.jses.2019.11.005. eCollection 2020 Mar. PMID 32195470
- [Background] Chau DL, Walker V, Pai L, Cho LM. Opiates and elderly: use and side effects. Clin Interv Aging. 2008;3(2):273-8. doi: 10.2147/cia.s1847. PMID 18686750
- [Background] Sabesan VJ, Chatha K, Koen S, Dawoud M, Gilot G. Innovative patient education and pain management protocols to achieve opioid-free shoulder arthroplasty. JSES Int. 2020 May 4;4(2):362-365. doi: 10.1016/j.jseint.2020.01.005. eCollection 2020 Jun. PMID 32490427
- [Background] Hasak JM, Roth Bettlach CL, Santosa KB, Larson EL, Stroud J, Mackinnon SE. Empowering Post-Surgical Patients to Improve Opioid Disposal: A Before and After Quality Improvement Study. J Am Coll Surg. 2018 Mar;226(3):235-240.e3. doi: 10.1016/j.jamcollsurg.2017.11.023. Epub 2018 Jan 10. PMID 29331347
- [Background] Nahhas CR, Hannon CP, Yang J, Gerlinger TL, Nam D, Della Valle CJ. Education Increases Disposal of Unused Opioids After Total Joint Arthroplasty: A Cluster-Randomized Controlled Trial. J Bone Joint Surg Am. 2020 Jun 3;102(11):953-960. doi: 10.2106/JBJS.19.01166. PMID 32251139
- [Background] Patel MS, Updegrove GF, Singh AM, Jamgochian GC, LoBiondo D, Abboud JA, Ramsey ML, Lazarus MD. Characterizing opioid consumption in the 30-day post-operative period following shoulder surgery: are we over prescribing? Phys Sportsmed. 2021 May;49(2):158-164. doi: 10.1080/00913847.2020.1789439. Epub 2020 Jul 9. PMID 32597282

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control/Standard of Care | Education Arm
Started | 68 | 72
Completed | 63 | 64
Not Completed | 5 | 8
Not completed — Surgery cancellation | 4 | 5
Not completed — didn't fill prescription | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control/Standard of Care | Education Arm | Total
Number analyzed (Participants) | 63 | 64 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.5) | 68.1 (7) | 67.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 29 | 52
  Male | 40 | 35 | 75
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Difference in Proportion of Participants With > 10 Pills Left Unused.
Description: Educational materials will be developed and their impact will be tested on opioid consumption patterns after total shoulder arthroplasty.
  By comparing Arm 1 and Arm 2 the investigators will determine the difference in opioid consumption between groups of patients who receive education and those who do not. Opioid consumption will be determined via patient self-reported opioid use on questionnaires completed during the first 2 weeks following surgery or at 6 weeks after surgery. The number of pills taken will be documented and will then be calculated by the research staff into MUE.
Time Frame: 2 weeks or 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control/Standard of Care | Education Arm
Number analyzed (Participants) | 63 | 64
Participants | 49 | 47

2. Secondary Outcome: Opioid Disposal
Description: Evaluate a structured and streamlined disposal protocol and its effect on opioid disposal rates.
  By comparing Arm 1 and Arm 2 the investigators will determine opioid disposal between subjects provided a structured disposal mechanism and those who are not provided a structured disposal mechanism. Opioid disposal will be measured via patient self-report. In each group participants will be asked how many pills were left unused and how many pills were disposed. This will be recorded on the postoperative surveys administered during the first 2 weeks following surgery, or at 6 weeks after surgery.
Time Frame: 2-weeks or 6-weeks post-operative.
Population: Percentage of participants who disposed unused opioid pills
Measure: Count of Participants; unit: Participants
Arm/Group | Control/Standard of Care | Education Arm
Number analyzed (Participants) | 60 | 59
Participants | 19 | 22

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control/Standard of Care | Education Arm
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/64
Other Adverse Events (participants affected / at risk) | 0/63 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT05525975/Prot_SAP_000.pdf